CLINICAL TRIAL: NCT02753985
Title: Adherence to Aromatase Inhibitors: The Role of Partners
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 15114
Record Dates: First submitted 2016-04-26; First posted 2016-04-28 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer Survivors
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Survey

SUMMARY:
This is a qualitative study which explores the role that partners play in breast cancer survivors adherence to aromatase inhibitors and management of their side effects. Both patients and their partners will be interviewed (separately) in order to capture multiple perspectives. The target number of subjects is 64 (32 patients and 32 partners). The primary method of data collection will be face-to-face semi-structured interviews. These interviews will be audio-recorded.

ELIGIBILITY:
Inclusion Criteria:

* Women and partners of women with stage I-III breast cancer who

  1. have completed primary cancer treatments (surgery, chemotherapy, radiotherapy)
  2. have experienced AI side effects
  3. live with a romantic partner.

     Exclusion Criteria:

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women and partners of women with stage I-III breast cancer
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-07; Primary Completion 2016-04-22 (Actual); Study Completion 2016-04-22 (Actual)

PRIMARY OUTCOMES:
Number of Surveys Completed | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun Mao, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States